CLINICAL TRIAL: NCT02437110
Title: HERV-K Suppression Using Antiretroviral Therapy in Volunteers With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150126; 15-N-0126
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2022-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Antiretroviral Therapy; Virus
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Virus Diseases | interventions — Darunavir; Ritonavir; dolutegravir; tenofovir alafenamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALS (Experimental): 20 participants with ALS and a level of HERV-K:RPP30 greater than or equal to 13
  Interventions: Drug: Darunavir; Drug: Ritonavir; Drug: Dolutegravir; Drug: Tenofovir alafenamide (TAF)

INTERVENTIONS:
Drug: Darunavir — Orally-administered medication approved for HIV treatment. MOA is as a protease inhibitor. Dose is 600mg twice daily.
Drug: Ritonavir — Orally-administered, FDA-approved medication for HIV treatment. Used in combination with darunavir. Dose is 100mg twice daily.
Drug: Dolutegravir — Orally-administered, FDA-approved medication to treat HIV. It acts as an integrase inhibitor. Dose is 50mg once daily.
Drug: Tenofovir alafenamide (TAF) — Orally-administered, FDA-approved medication used to treat HIV. It acts as a nucleoside reverse transcriptase inhibitor. Dose is 25mg once daily.

SUMMARY:
Background:

Some people with Amyotrophic Lateral Sclerosis (ALS) have a high level of the virus HERV-K in their blood. Researchers do not think this virus causes ALS. But they don t know why some people with ALS have a high level of it. They want to know if HERV-K can be suppressed by drugs that are used to treat HIV infection.

Objectives:

To learn how drugs usually taken for HIV infection affect people with Amyotrophic Lateral Sclerosis (ALS).

Eligibility:

Adults at least 18 years old with ALS and high levels of HERV-K but no HIV.

Design:

Interested participants can contact the study team and, if eligible, the study team will arrange for a screening blood draw to determine the HERV-K level.

Participants with a high HERV-K level will be screened with medical history, physical exam, questionnaires, nerve conduction test, lumbar puncture, and blood and breathing tests.

After screening, participants will start taking the 4 study drugs.

Participants will have up to 12 study visits over a period of 72 weeks. After starting study drugs, they will have study visits at Weeks 1 and 4 and then every 4 weeks until Week 28. They will be asked how they are feeling and have an exam and blood drawn. At 3 visits, they will have tests of nerve conduction, breathing, and their ALS symptoms.

At Week 24, they will stop taking the study drugs and may have a repeat lumbar puncture.

After the Week 48 visit, their participation is finished.

DETAILED DESCRIPTION:
Objective:

In this Phase I, proof-of-concept study, we aim to determine whether an antiretroviral regimen approved to treat human immunodeficiency virus (HIV) infection would also suppress levels of Human Endogenous Retrovirus-K (HERV-K) found to be activated in a subset of patients with amyotrophic lateral sclerosis (ALS). We propose to measure the blood levels of HERV-K before, during, and after treatment with an antiretroviral regimen. We will evaluate the safety of the antiretroviral regimen for participants with ALS and also explore clinical and neurophysiological outcomes of ALS symptoms, quality of life, and pulmonary function.

Study Population:

We will study a subset of ALS patients who have a ratio of HERV-K:RPP30 greater than or equal to 13. About 30% of ALS patients may have detectable levels of HERV-K; about 20% of patients with ALS have a level >1000 copies/ml. To show whether the HERV-K could be suppressed, we will recruit from the approximately 20% of patients with high levels so that the antiretroviral effect can be determined.

Design:

This is an open-label study of a combination antiretroviral therapy for 24 weeks in 25 HIV-negative, HTLV-negative ALS patients with high ratio of HERV-K:RPP30. The study duration for each participant will be up to 72 weeks. Participants will be followed regularly for safety, clinical, and neurophysiological outcomes.

Outcome Measures:

The primary outcome measure will be the percent decline in HERV-K concentration. Percent decline for a patient is measured by: 100 x (screening visit - week 24 visit measurement) / screening visit. The safety of antiretrovirals in volunteers with ALS as measured by the frequency and type of AEs, the ability to remain on assigned treatment (tolerability), physical examinations, laboratory test results, vital signs, and weight. Efficacy will be explored by measuring the change in mean scores of: the ALS Functional Rating Scale-Revised (ALSFRS-R), the ALS Specific Quality of Life Inventory-Revised (ALSSQOL-R), the ALS Cognitive Behavioral Screen (ALS-CBS), vital capacity and maximal inspiratory pressure as measured by handheld spirometer, electrical impedance myography (EIM), the change in neurofilament levels in blood and/or CSF, and the change in urine p75ECD levels.

ELIGIBILITY:
INCLUSION CRITERIA:

Subjects must meet all of the following inclusion criteria to be eligible to participate in this study:

Age 18 years or older at the time of the screening visit.

Able to provide informed consent and comply with study procedures.

ALS diagnosed as probable, laboratory-supported probable or definite according to the World Federation of Neurology El Escorial revised criteria as determined by a neurologist with neuromuscular subspecialty training.

A ratio of HERV-K:RPP greater than or equal to 13 measured by quantitative PCR at the screening visit.

Duration of disease less than 2 years, or if greater than 2 years, disease progression at a rate that in the judgement of the investigator would allow for completion of the study.

If taking riluzole or edaravone, must be on a stable dose for at least 30 days prior to the screening visit, or stopped taking riluzole or edaravone at least 30 days prior to the screening visit.

Subject has a competent caregiver who can and will be responsible for administering study drug. If there is no caregiver, another qualified individual must be available to do this.

Subject has established care with a neurologist and will maintain this clinical care throughout the study.

Subject has had neuroimaging within the last 24 months for participants enrolling at the NIH Clinical Center.

EXCLUSION CRITERIA:

A participant will be excluded if he or she has any of the following:

Dependence on daytime mechanical ventilation (invasive or non-invasive, including Continuous Positive Airway Pressure (CPAP) or Bilevel Positive Airway Pressure (BiPap) at the time of the screening visit.

Participation in any other investigational drug trial or using investigational drug (within 4 weeks prior to the Day 0 visit and thereafter).

History of severe sulfonamide allergy (i.e. anaphylaxis).

History of positive test or positive result at screening for HIV or HTLV-1.

Participants must not be able to become pregnant (e.g., post-menopausal for at least one year, surgically sterile, or using adequate methods of contraception) or breastfeed for the duration of the study. Adequate methods of contraception include: implanted contraception, intrauterine device in place for at least 3 months, or barrier method in conjunction with spermicide. Participants of childbearing potential must have a negative pregnancy test at screening and be non-lactating.

Presence of any of the following clinical conditions at the time of screening:

Drug abuse or alcoholism

Unstable medical disease (such as unstable angina or chronic obstructive pulmonary disease), or active infectious disease (such as Hepatitis C or tuberculosis), or current malignancy

Unstable psychiatric illness defined as psychosis or untreated major depression within 90 days of the screening visit

Dementia

Diabetes mellitus

Hemophilia

Use of contraindicated medications: amiodarone, dronedarone, lovastatin, simvastatin, rifampin, rifapentine, rifabutin, cisapride, pimozide, midazolam, triazolam, dihydroergotamine, ergonovine, ergotamine, methylergonovine, St. John s wort, alfuzosin, salmeterol, sildenafil for pulmonary arterial hypertension, oxcarbazepine, phenobarbital, phenytoin or dofetilide.

Safety Laboratory Criteria at the screening visit:

Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 3.0 times the upper limit of normal

Serum creatinine, serum phosphorous, total bilirubin, triglycerides, amylase, or lipase greater than 2.0 times the upper limit of normal

Estimated glomerular filtration rate <60mg/dl.

Platelet concentration of <100,000/ (micro)l.

PT and PTT >1.2 times the upper limit of normal for participants enrolling at the NIH Clinical Center.

Hemoglobin <10mg/dL.

Positive Hepatitis B Surface Antigen and Hepatitis C Virus Antigen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2023-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avindra Nath, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andrews WD, Tuke PW, Al-Chalabi A, Gaudin P, Ijaz S, Parton MJ, Garson JA. Detection of reverse transcriptase activity in the serum of patients with motor neurone disease. J Med Virol. 2000 Aug;61(4):527-32. doi: 10.1002/1096-9071(200008)61:43.0.co;2-a. PMID 10897073
- [Background] Douville R, Liu J, Rothstein J, Nath A. Identification of active loci of a human endogenous retrovirus in neurons of patients with amyotrophic lateral sclerosis. Ann Neurol. 2011 Jan;69(1):141-51. doi: 10.1002/ana.22149. PMID 21280084
- [Background] Moulignier A, Moulonguet A, Pialoux G, Rozenbaum W. Reversible ALS-like disorder in HIV infection. Neurology. 2001 Sep 25;57(6):995-1001. doi: 10.1212/wnl.57.6.995. PMID 11571323
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-N-0126.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were referred to the study by their provider or self-referred between April 2019 and June 2022. In total,122 participants were screened to determine HERV-K levels and eligibility to the treatment arm of the study. 118 participants were screened in protocol 15N0126 (Period 1) and 4 were screened in a companion protocol.
Pre-assignment Details: 34 participants qualified and were interested in participating in the treatment portion of the protocol (Period 2). The follow-up period (Period 3), included a post treatment follow-up period from week 24 to week 48. Of the 20 participants who completed the treatment portion of the protocol,19 qualified for the follow-up period. One participant was excluded from the follow-up period (Period 3) due to a deviation from the protocol.
Groups:
- Participants With ALS: Adults with sporadic or familial ALS
Period: Screening
Arm/Group | Participants With ALS
Started | 118
Completed | 114
Not Completed | 4
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 1
Period: ART
Arm/Group | Participants With ALS
Started | 34
Completed | 20
Not Completed | 14
Not completed — Adverse Event | 3
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 4
Not completed — Lost to follow-up prior to start of intervention | 1
Not completed — Physician decision prior to start of intervention | 2
Not completed — Withdrawal by subject prior to starting intervention | 1
Period: Post-ART
Arm/Group | Participants With ALS
Started | 19
Completed | 9
Not Completed | 10
Not completed — Lost to Follow-up | 3
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Represents those participants receiving the study intervention, i.e., antiretroviral treatment.
Groups:
- ALS ART Treatment: Participants with ALS participating in the treatment period of the trial.
Arm/Group | ALS ART Treatment
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in HERV-K Level
Description: Blood samples were obtained during the screening visit and week 24 (post-treatment with antiretroviral drugs). The percent change in HERV-K level was measured using quantitative PCR: 100% x (screening visit - week 24 visit measurement) / screening visit.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: Percent change
Groups:
- Patients With HERV-K 13: 20 participants with ALS and a level of HERV-K:RPP30 greater than or equal to 13
Arm/Group | Patients With HERV-K 13
Number analyzed (Participants) | 20
Percent change | -30.7 (0.06)

ADVERSE EVENTS:
Time Frame: 48 weeks
Groups:
- Screening Period: Adverse events noted in participants during the Screening period
- ART Treatment Period: Adverse events noted in participants during the ART Treatment period
- Post-ART Follow-Up Period: Adverse events noted in participants following the ART Treatment period
Arm/Group | Screening Period | ART Treatment Period | Post-ART Follow-Up Period
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/34 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/118 | 0/34 | 0/19
Other Adverse Events (participants affected / at risk) | 0/118 | 30/34 | 3/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screening Period (N=118) | ART Treatment Period (N=34) | Post-ART Follow-Up Period (N=19)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 8 (8) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Blood Bicarbonate Decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Cerebrospinal Fluid Leakage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cholesterol High (Investigations) | 0 (0) | 14 (14) | 0 (0)
CPK Increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Creatinine Increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 8 (8) | 0 (0)
Gastrointestinal Disorders - other, bowel urgency (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Disorders - other, large bowel movement (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Glucose Intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 11 (11) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 11 (11) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 11 (11) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Lipase Increased (Investigations) | 0 (0) | 3 (3) | 1 (1)
Localized Edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 6 (6) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Serum Amylase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT02437110/Prot_SAP_001.pdf
  • Informed Consent Form (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT02437110/ICF_002.pdf